CLINICAL TRIAL: NCT02504112
Title: Evaluation of Zimmer® CAS PSI X-Ray Knee in Total Knee Arthroplasty (TKA): Technical Outcomes
Brief Title: Zimmer CAS PSI X-Ray Knee in TKA (Total Knee Arthroplasty)
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSU2015-12K
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Total Knee Arthroplasty / Position of Customized X-Ray PSI Guides Using Optical Navigation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- X-Ray PSI Group: Male or female patients, over 18 years old and with indication of total knee arthroplasty
  Interventions: Other: there is no intervention

INTERVENTIONS:
Other: there is no intervention

SUMMARY:
The objective of the observational study is to assess the positioning of customized guides designed from patients X-Rays (Zimmer® X-Ray PSI Knee) using optical navigation in primary total knee arthroplasty.

DETAILED DESCRIPTION:
The proposed research is a single center, prospective, case series, and non-controlled study. One orthopedic surgeon will perform 30 primary TKAs using X-Ray PSI Knee guides, generated from X-ray. Patients who have been appropriately indicated as candidates for TKA and who meet the specified inclusion and exclusion criteria, will be informed about Zimmer® X-Ray PSI Knee technology and offered entry into the study. Informed consent, in accordance with current ethical board regulatory requirements and best practice, will be obtained from all patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Needs a primary TKA and he/she is Persona® knee implant compatible
* Diagnosed with non-inflammatory degenerative joint disease (e.g., osteoarthritis, post-traumatic arthritis, avascular necrosis, etc.)
* Over 18 years old
* Able to:
* Understand what participation in the study entails and willing to consent (patient or his/her legal guardian) to participate in the study by signing and dating an IRB/EC approved inform consent form. and
* Follow surgeon/staff instructions, and
* Return for all follow-up evaluations, and
* Able and willing to undergo a preoperative radiographs (all cases)
* Meets an acceptable preoperative medical clearance and is free of or treated for cardiac, pulmonary, hematological or other conditions that would pose excessive operative risk.
* Has a presence of varus or valgus deformity of 15 degrees or less.

Exclusion Criteria:

* Is currently enrolled in an investigational new drug or device study
* Has an active infection (including septic knee, distant infection, or osteomyelitis)
* Has neurological disorders (including, but not limited to Parkinson's disease)
* Has had a prior ipsilateral unicompartmental knee arthroplasty, TKA, knee fusion or patellectomy.
* Has hip or knee ankylosis.
* Have indications of intra- and/or extra-articular deformations that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately sized implant, such as polio, history of tibial plateau fracture, etc.
* Has any metal within 150 mm of the joint line for the operative-side knee.
* Has knee deformities greater than 15 degrees of fixed varus, valgus, or flexion contracture on initial physical examination.
* Is a female who is pregnant or lactating
* Is currently involvement in any personal injury litigation, medical-legal or worker's compensation claims
* Has arterial disease or stents that would exclude the use of a tourniquet.
* Has insufficient quality or quantity of bone to support the implant due to prior knee surgery (or surgeries), cancer, metabolic bone disease, osteoporosis/osteopnea (diagnosed or treated with medication), active/old/remote infection, etc.
* Has a mental condition that may interfere with his/her ability to give an informed consent or interfere with his/her ability or willingness to fulfill the requirements of the study.
* Has a condition that would place excessive demands on the implant (e.g., Charcot's joints, muscle deficiencies, multiple joint disabilities, skeletal immaturity, etc.).
* Has collateral ligament insufficiency.
* Has an immunosuppressive disorder (e.g., AIDS, etc.) that would require cytotoxic drugs, corticosteroids, large dose of irradiation, or antilymphocytic serum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with indication of Total Knee Arhtroplasty
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
assess the positioning accuracy and precision of customized X-RAY PSI guides using the Sesamoid Optical Navigation system in Total Knee Arthroplasty | Intra-operative

SECONDARY OUTCOMES:
assess the correlation between planned vs. actual component size and bony resection thickness | Intra-operative